CLINICAL TRIAL: NCT00325507
Title: Safety, Immunology, and Biological Activity Evaluation of TroVax® in Treatment of Patients With Locally Advanced or Metastatic Renal Carcinoma
Brief Title: Safety and Biological Activity of TroVax® Vaccine Given With IL-2 in Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford BioMedica (Industry)
Collaborators: The Methodist Hospital Research Institute (Other); ORION Clinical Services (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV-B2/001/05
Record Dates: First submitted 2006-05-10; First posted 2006-05-12 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Carcinoma, Renal Cell
Keywords: renal cell carcinoma; requiring IL-2 treatment; Locally advanced or metastatic renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — TroVax; Interleukin-2

ARMS (1):
- TroVax (Experimental): TroVax given as first or second line treatment in conjuntion with low dose IL-2.
  Interventions: Biological: TroVax; Drug: IL-2

INTERVENTIONS:
Biological: TroVax — TroVax 1 x 10E9 TCID 50mL
Drug: IL-2 — IL-2 250,000 U/kg S/C for cycle 1 and day 1 of subsequent cycles, 125,000U/kg S/C for days 2-5 of cycles 2-6

SUMMARY:
The purpose of this study is to assess the safety and tolerability of TroVax® investigational vaccine injections when given as first or second line treatment in conjunction with subcutaneous low dose IL-2 to patients with locally advanced or metastatic clear cell or papillary cell renal carcinoma.

TroVax® is the experimental product in this trial and its value as a medicine has not yet been proven. Interleukin-2 (IL-2) is a standard treatment for cancer, which means that it can be received even if one chooses not to participate in this study. TroVax® is being studied as a possible treatment for patients with cancer of the kidney.

TroVax® belongs to a class of medicines called vaccines. A vaccine helps the body's immune system to recognize and kill foreign invading organisms effectively. It is believed that one of the reasons why cancer can spread through the body is that the immune system cannot recognize cancer cells as being different from normal tissues and therefore cannot kill the cancer cells. A vaccine that alerts the immune system to the presence of cancer cells in the body could lead to the immune system being able to target and kill those cancer cells effectively. This trial is of a completely new way of trying to treat cancer in the future by the use of vaccination injections. TroVax® consists of a virus that has been changed so that it is no longer infectious and carries a gene for a protein called 5T4. This protein is carried by many kidney cancer cells. When the virus is injected, it makes the protein, and the body's immune system is then able to recognize this protein and kill the cells that have it (i.e. the cancer cells).

The purpose of this study is to assess the safety and tolerability of TroVax® injections and to understand whether TroVax® could make such an immune response happen in patients with renal cell cancer while receiving interleukin-2 (IL-2). This study will also observe and monitor any side effects experienced in patients who receive TroVax® while being treated with IL-2.

DETAILED DESCRIPTION:
Objectives

Primary:

* To assess the safety and tolerability of TroVax® injections when given as first or second line treatment in conjunction with subcutaneous low dose IL-2 to patients with locally advanced or metastatic clear cell or papillary cell renal carcinoma.
* To assess the immune responses induced by treatment with TroVax® and subcutaneous low dose IL-2.

Secondary:

* To assess tumour response rates, time to progression, survival and progression free survival at 6, 12 and 24 months after commencement of treatment with subcutaneous low dose IL-2.
* To assess the ability of the reintroduction of low dose subcutaneous IL-2 to induce further disease responses or stabilisation in patients being treated with TroVax® alone.

Study design:

This will be an open label evaluation in patients with clear cell or papillary cell renal carcinoma requiring immunotherapy for locally advanced or metastatic disease. A single dose level of TroVax® in combination with a clinically accepted regimen of subcutaneous low dose IL-2 will be tested in 25 evaluable patients and their immunological responses to TroVax® (antibody and cellular) will be assessed. If immunological activity is observed after two cycles of TroVax®/IL-2 in 70% or more of these patients, further randomised trials will be undertaken to determine the clinical efficacy of TroVax® in this group of patients.

The dosage schedule of subcutaneous low dose IL-2 will be an initial dose schedule of 250,000 U/kg/dose for 5 days in week 1 followed by 125,000 U/kg/dose for 5 days in each of weeks 2 though 6 inclusive. There will then be a two-week recovery period before the next cycle commences. The dosage regimen of TroVax® will be injections given prior to the first cycle on two occasions (weeks -2 and 1), and one injection given at the beginning of week 4 of the first cycle. In subsequent cycles, booster injections of TroVax® will be given at week 1 only, prior to commencement of subcutaneous IL-2 therapy. After the first and second cycles of combined treatment, patients will be evaluated by CT scan for their response to treatment. If their disease has progressed after the second cycle, they will be withdrawn from the trial if they require alternative therapy (deterioration of one level of the Karnofsky score or appearance of disease in a new site). If they are experiencing progressive disease that does not require alternative therapy or stable disease or better, they will be treated with cycles of TroVax®/IL-2 as described above for up to a further four cycles. The tumour status will be evaluated by CT scan after every cycle.

All patients will be monitored for up to 6 cycles (48 weeks) to assess tolerability, induction of humoural and cellular immunity to 5T4 cell surface antigen, immune response to the vector, tumour response rates, survival, time to progression and progression free survival. Patients who are intolerant of further treatments with subcutaneous IL-2 during this part of the study will be withdrawn from the study.

Patients who are still stable or experiencing a tumour response at 48 weeks will be offered further boosts with TroVax® without IL-2 every three months at weeks 52, 64, 76, 88 and 100. During this period, if disease progression recurs, two further cycles with subcutaneous IL-2 as described above may be given in combination with TroVax® as described above with the objective of inducing further disease response or stabilisation.

Following termination of all patients' participation in the trial (including those with progressive disease after two cycles of TroVax®/IL-2), contact will be kept by the Investigators with their families in order to determine the date of death.

A total of 25 patients will be enrolled.

Withdrawal criteria from the trial:

1. Non-compliance with the protocol.
2. Patient withdraws consent.
3. Progressive disease with new sites of disease demonstrated on CT scan and/or requiring other cancer treatment (deterioration in Karnofsky performance score of 10% or more).
4. Death.
5. Serious IL-2 related adverse events or lack of tolerance to further treatment with IL-2
6. Serious TroVax® related adverse events (DLT).

   Treatment plan and methods:

   Patients complying with the entry criteria will be invited to enter the study. After giving fully informed consent, patients will be subjected to a physical examination to document general fitness to proceed with the trial. Vital signs will be recorded. Performance status (Karnofsky) will be documented. At that time, metastases will be documented using chest, abdominal and pelvic CT scans and an MRI scan of the brain will be obtained. Blood samples will also be obtained for clinical pathology (10 mL; safety testing). A urine sample will be tested for protein and blood (safety testing). A 12 lead ECG and echocardiogram will be obtained. This screen should not occur more than two weeks before treatment with TroVax® begins. If available, tumour tissue from earlier biopsies will be obtained and tested for the presence of tumour antigens, e.g. 5T4. CT scans must be compared with scans obtained within the previous three months in order to determine that the disease is progressing.

   Week -2, day 1:

   Obtain blood sample for HLA testing and immunological evaluation, (antibody and T-cell responses to the vector and the 5T4 surface antigen; 100 mL).

   Safety testing (blood, 10 mL and urine) TroVax® injection i.m. 1 mL

   Cycle 1, Week 1 day 1:

   Karnofsky score Vital signs TroVax® injection i.m. 1 mL (time 0) Vital signs (1 hour) / Vital signs (3 hours) IL-2 subcutaneous injection (250,000 U/kg/dose) safety testing

   Cycle 1, Week 1, days 2-5:

   IL-2 subcutaneous injection (250,000 U/kg/dose)

   Cycle 1, Week 2, day 1:

   Obtain samples for immunological evaluation (100 mL blood) and safety testing (blood 10 mL and urine) IL-2 subcutaneous injection (125,000 U/kg/dose).

   Week 2, days 2-5:

   IL-2 injection subcutaneous (125,000 U/kg/dose).

   Week 3, days 1-5:

   Safety testing (blood and urine; day 1 only) IL-2 subcutaneous injection (125,000 U/kg/dose).

   Week 4, day 1:

   Safety testing Vital signs TroVax® injection i.m. 1 mL (time 0) Vital signs (1 hour) / Vital signs (3 hours) IL-2 subcutaneous injection (125,000 U/kg/dose).

   Week 4, days 2-5:

   IL-2 subcutaneous injection (125,000 U/kg/dose).

   Week 5, days 1-5:

   Obtain sample for immunological evaluation (blood) and safety testing (blood 10 mL and urine; day 1 only) IL-2 subcutaneous injection (125,000 U/kg/dose).

   Week 6, days 1-5:

   Obtain sample for safety testing (blood 10 mL and urine; day 1 only) IL-2 subcutaneous injection (125,000 U/kg/dose).

   Week 8 day 1:

   CT scan for information. Physician examination. Safety blood (10 mL) and urine

   Cycles 2-6 week 1, day 1:

   Obtain sample for safety testing (blood 100 mL and urine) Vital signs Karnofsky score TroVax® injection i.m. 1 mL (time 0) Vital signs (1 hour) / Vital signs (3 hours) IL-2 subcutaneous injection (250,000 U/kg/dose)

   Cycle 2-6, week 1, days 2-5:

   IL-2 subcutaneous injection (250,000 U/kg/dose)

   Cycles 2-6, Week 2, day 1:

   Obtain sample for immunological evaluation (blood) and safety testing (blood and urine).

   IL-2 subcutaneous injection (125,000 U/kg/dose).

   Cycles 2-6, Week 2, days 2-5:

   IL-2 subcutaneous injection (125,000 U/kg/dose).

   Cycles 2-6, Weeks 3-6, days 1-5:

   Safety testing (blood 10 mL and urine day 1 only) IL-2 subcutaneous injection (125,000 U/kg/dose)

   Cycles 2-6, Week 8, day 1:

   Obtain blood for safety testing (blood and urine) CT scan. Physician examination.

   At the end of cycle 2 to 6 inclusive, if disease has progressed and requires other treatment (deterioration in Karnofsky performance score by 10% or more, disease appears in a new site), withdraw patient from trial. Also withdraw patient if intolerant of subcutaneous low dose IL-2 at the lowest permissible dose or if the patient experiences DLT. Patients withdrawing before they receive the first four doses of TroVax® and give blood for immunology testing in cycle 2, week 2 will be replaced.

   If disease is stable, responding or progressing (but Karnofsky score unchanged, no new disease sites) and patient is tolerant of treatment, continue with further therapy.

   After six cycles of combined study drugs (48 weeks), assess with CT scan at week 48 day 1:

   If disease has progressed and requires alternative treatment (deterioration in Karnofsky performance score by 10% or more or disease appears in a new site), withdraw patient from trial.

   If disease is stable or responding or progressing (but Karnofsky score stable and no new disease sites) and patient is tolerant of treatment, continue with further therapy. This therapy will be TroVax® injection every three months, on weeks 52, 64, 76, 88, 100. Perform physician examination on each occasion and assess Karnofsky score prior to injection. Obtain samples for safety testing (blood 10 mL and urine) and immunological evaluation (10 mL sample only for antibody testing) prior to each injection. A further 10 mL sample for immunological evaluation will be obtained one week after each TroVax® injection. CT scans will be obtained at weeks 63, 75, 87, 99. At each CT scan, assess:

   If disease has progressed, recommence subcutaneous low dose IL-2 treatment (6 weeks on, two weeks off IL-2) at week 64, 76, 88 as appropriate and give a further 2 cycles of subcutaneous low dose IL-2.

   If IL-2 restarted at week 64 (76, 88), schedule is:

   Week 64 (or 76, 88), day 1:

   Safety testing (blood 10 mL and urine) TroVax® injection i.m. 1 mL Karnofsky score IL-2 subcutaneous injection (250,000 U/kg/dose) Physical examination

   Week 64 (or 76, 88), days 2-5:

   IL-2 subcutaneous injection (250,000 U/kg/dose)

   Week 65 (or 77, 89), days 1-5:

   Safety testing (blood 10 mL and urine, day 1 only). Immunological evaluation, 10 mL sample only (day 1 only) IL-2 subcutaneous injection (125,000 U/kg/dose).

   Weeks 66-69 (or 78-81, or 90-93), days 1-5:

   Safety testing (blood 10 mL and urine, day 1 only). IL-2 subcutaneous injection (125,000 U/kg/dose).

   Week 71 (or 83 or 95) day 1:

   Physician examination. CT scan.

   Second Cycle:

   Week 72 (or 84, 96), day 1:

   Safety testing (blood 10 mL and urine) TroVax® injection i.m. 1 mL Karnofsky score IL-2 injection (250,000 U/kg/dose)

   Week 72 (or 84, 96), days 2-5:

   IL-2 injection (250,000 U/kg/dose)

   Week 73 (or 85, 97), days 1-5:

   Safety testing (blood 10 mL and urine, day 1 only). Immunological evaluation, 10 mL sample only (day 1 only) IL-2 subcutaneous injection (125,000 U/kg/dose).

   Weeks 74-77 (or 86-89, or 98-101), days 1-5:

   Safety testing (blood and urine, day 1 only). IL-2 subcutaneous injection (125,000 U/kg/dose).

   Week 79 (or 91 or 103) day 1:

   Physician examination. CT scan.

   After the second cycle of IL-2, if disease has progressed and requires other treatment (deterioration in Karnofsky score by 10% or more, disease appears in a new site), withdraw patient from trial.

   If the treatment cycles with IL-2 end before week 104 and the patient is responding, stable or progressing but not in need of alternative therapies (Karnofsky stable, no new disease sites), recommence TroVax® on the original schedule (see Flow Chart). If disease is progressing and requires further therapy (deterioration in Karnofsky score by 10% or more, disease appears in a new site), withdraw patient from trial.

   Four weeks after the final treatment, all patients will, if possible, attend for a final follow up visit. The following will be obtained:

   Physical examination. Karnofsky score Safety testing (blood 10 mL and urine).

   All study visits must occur within +/- 3 days of the day stipulated in the protocol.

   If patients withdraw at any time during the trial, a final follow up visit, if possible, will be obtained four weeks after withdrawal.

   Concomitant medication and adverse events will be recorded at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced or metastatic, histologically proven clear cell or papillary cell renal carcinoma.
2. Primary tumour surgically removed.
3. Progressive disease
4. At least four weeks from any previous therapy for renal cancer.
5. Fit for first or second line immunotherapy with subcutaneous low dose IL-2
6. Measurable disease
7. Aged 18 years or more.
8. Patients must comply with the following:

   * Karnofsky score ≥ 80%
   * Corrected calcium ≥ 10 g/dL (2.5 mmols/L)
9. Clinically immunocompetent
10. Free of clinically apparent autoimmune disease.
11. Haemoglobin ≥ 9 g/dL, total white cell count ≥ 3 x 10^9/L and lymphocyte count ≥ 1 x 10^9/dL
12. Serum creatinine up to 1.5 times upper limit of normal.
13. Bilirubin ≤ 2 mg% and an SGPT of ≤ 4 times the upper limit of normal.
14. Able to give written informed consent and to comply with the protocol.
15. Women must be either post menopausal, or rendered surgically sterile or, if of child bearing potential, must have been practising a reliable form of contraception (oral contraception + a barrier method) for at least three months prior to the first dose of TroVax® and must continue while they are being treated with TroVax®. Men must practise a reliable form of contraception while they are being treated with TroVax®.
16. No acute changes on 12-lead electrocardiogram (ECG)
17. Ejection fraction on echocardiogram ≥ 45%

Exclusion Criteria:

1. Previous immunotherapy with any schedule of IL-2.
2. Intercurrent serious infections within the 28 days prior to entry into the trial.
3. Life threatening illness unrelated to cancer.
4. Cerebral metastases on MRI scan.
5. History of allergic response to previous vaccinia vaccinations.
6. Participation in any other clinical trial of a licensed or unlicensed drug within the previous 30 days or during the course of this trial.
7. Previous malignancies within the last 10 years other than successfully treated squamous carcinoma of the skin or in situ carcinoma of the cervix treated with cone biopsy.
8. Previous history of major psychiatric disorder requiring hospitalisation or any current psychiatric disorder that would impede the patient's ability to provide informed consent or to comply with the protocol.
9. Known allergy to egg proteins
10. Chronic oral corticosteroid use unless prescribed as replacement therapy in the case of adrenal insufficiency.
11. Known to test positive for HIV or hepatitis B or C
12. Known hypersensitivity to neomycin
13. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TroVax injections in conjunction with low dose IL-2 | 48 weeks
  To assess the safety and tolerability of TroVax injections when given as first or second line treatment in conjunction with subcutaneous low dose IL-2 to patients with locally advanced or metastatic clear cell or papillary cell renal carcinoma.
  To assess the immune responses induced by treatment with TroVax and subcutaneous IL-2

SECONDARY OUTCOMES:
Tumour Response Rates | 6, 12 & 24 months
  To assess tumour response rates, time to progression, surgival and progression free surgival at 6, 12 and 24 months after commencement of treatment with subcutaneous low dose IL-2.
  To assess the ability of the reintroduction of low dose subcutaneous IL-2 to induce further disease responses or stabilisation in patients being treated with TroVax alone.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Amato RJ, Shingler W, Naylor S, Jac J, Willis J, Saxena S, Hernandez-McClain J, Harrop R. Vaccination of renal cell cancer patients with modified vaccinia ankara delivering tumor antigen 5T4 (TroVax) administered with interleukin 2: a phase II trial. Clin Cancer Res. 2008 Nov 15;14(22):7504-10. doi: 10.1158/1078-0432.CCR-08-0668. PMID 19010868